CLINICAL TRIAL: NCT01651832
Title: Supportive Cancer Care Networkers - a Prospective Randomized Controlled Multi-center Trial
Brief Title: Supportive Cancer Care Networkers (SCAN)
Acronym: SCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Alexander Bauer, Scientific Research Fellow, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01GY1143
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer; Chemotherapy
Keywords: Colorectal Neoplasms/*drug therapy/*secondary; Health Services Accessibility; Humans; Supportive Care Needs; Psychooncology; Rural Population; Primary Health Care/*methods; Treatment Outcome; Socioeconomic Factors; Quality Assurance, Health Care; Quality of Life; Adult; Aged; Aged, 80 and over
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention): routine care and case management
- SCAN-Intervention (Experimental)
  Interventions: Behavioral: SCAN

INTERVENTIONS:
Behavioral: SCAN — The Supportive Cancer Care Networkers intervention (SCAN) consists of an additional telephone support and symptom-related out-patient care management through Oncology Nursing. The SCAN intervention assesses patients' resources and barriers in utilizing health care services in order to meet their individual needs adequately and supports maintenance of therapy compliance. Thus, the SCAN offers a comprehensive mirroring the patients' medical and psychosocial care needs across changing sectors of health care.
  Arms: SCAN-Intervention

SUMMARY:
Aim of the study is to increase the proportion of indicated patients with colorectal cancer undergoing adjuvant chemotherapy following surgical resection through an optimized symptom management and logistical support.

DETAILED DESCRIPTION:
Patients with colorectal cancer in Germany today are exposed to several Problems related to care continuity and access to health care professionals. In order to increase the utilization of adjuvant therapies, patients in the intervention group are offered an additional nursing intervention in the period between discharge after inpatient treatment and the beginning of adjuvant therapy. This includes a telephone follow-up conducted according to guidelines serving to disclose patients' current supportive needs in order to determine potential intervention approaches as early as possible. Hence, the intervention aims to motivate patients not to discontinue the treatment. An early detection of therapy-related physical and psychological impairments aims at optimizing treatment management.

Patients in the intervention group therefore are visited by nursing staff specialized in cancer care (Supportive Cancer Care Networkers, SCAN) during their in-patient stay and are informed about the intervention. An assignment for the SCAN is to support patients in getting access to health care services (e.g. specialists). Patients are given certain information, as for example contact to specialists, voluntary services and the next steps and appointments of the treatment plan are discussed. Within a consultation at the day before hospital discharge, the SCAN takes up the contact information and appoints weekly telephone consultations for the time up to the adjuvant therapy. The SCAN hands out information materials and explains the study documents, as for example patient-held records (PHR) in order to improve therapy compliance.

ELIGIBILITY:
Inclusion Criteria:

* colorectal carcinoma (ICD-10: C18, C19, C20)
* indication for adjuvant chemo therapy following S3-Guideline on colorectal Cancer or physician-directed
* living in Saxony-Anhalt
* ECOG-Performance Status <3
* prospective further life expectancy of more than three months

Exclusion Criteria:

* unable to read or understand German properly
* any contra-indication for adjuvant therapy as described in the S3-Guideline such as inadequate liver, bone marrow, and kidney function or coronary heart disease (NYHA III-IV).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
proportion of eligible patients undergoing adjuvant chemo therapy | 8 weeks after hospital discharge/ chrirurgical resection

SECONDARY OUTCOMES:
disease-free survival | 8 month after hospital discharge/ chrirurgical resection
Health-related Quality of Life | 8 weeks & 8 month after hospital discharge/ chrirurgical resection
  using the EORTC QLQ-C30 & CR-29
symptom burden | 8 weeks & 8 month after hospital discharge/ chrirurgical resection
  using the M.D. Anderson Symptom inventory
Distress | 8 weeks & 8 month after hospital discharge/ chrirurgical resection
  using the Distress-Thermometer
supportive care needs | 8 weeks & 8 month after hospital discharge/ chrirurgical resection
  using the Supportive Needs Questionnaire-37 (FU-T)
Quality of inpatient care | at Baseline
  using the EORTC INPATSAT-32

CONTACTS AND LOCATIONS:
Overall Officials: Margarete Landenberger, Prof. Dr., Study Director — Martin-Luther-University Halle-Wittenberg, Medical Faculty, Institute for Health and Nursing Science
Locations (9):
- Germany (9):
  - Diakonissen-Krankhenhaus Leipzig, Leipzig, Saxony
  - AMEOS Klinikum Aschersleben-Staßfurt GmbH, Aschersleben, Saxony-Anhalt
  - Diakonissenkrankenhaus Dessau gGmbH, Dessau, Saxony-Anhalt
  - HELIOS Klinik Lutherstadt Eisleben, Eisleben Lutherstadt, Saxony-Anhalt
  - University Hospital Halle, Halle, Saxony-Anhalt
  - Klinikum Magdeburg gGmbH, Magdeburg, Saxony-Anhalt
  - HELIOS Klinik Sangerhausen, Sangerhausen, Saxony-Anhalt
  - AMEOS Klinikum Schönebeck GmbH, Schönebeck, Saxony-Anhalt
  - Carl-von-Basedow-Klinikum Merseburg, Merseburg, Saxony-Anhat

REFERENCES:
- [Derived] Bauer A, Vordermark D, Seufferlein T, Schmoll HJ, Dralle H, Mau W, Unverzagt S, Boese S, Fach EM, Landenberger M. Trans-sectoral care in patients with colorectal cancer: Protocol of the randomized controlled multi-center trial Supportive Cancer Care Networkers (SCAN). BMC Cancer. 2015 Dec 22;15:997. doi: 10.1186/s12885-015-2002-6. PMID 26694748